CLINICAL TRIAL: NCT01920516
Title: Prospective Observational Study on Isolated Limb Perfusion of Melphalan in Treating Patients With Metastasis or Recidivism of Limb Melanoma or Sarcoma That Are Not Operable
Brief Title: Isolated Limb Perfusion of Melphalan for Melanoma and Sarcoma Treatment
Acronym: ILI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Group of Endovascular Oncology (Other)
Responsible Party: Principal Investigator, Giammaria Fiorentini, Dr., International Group of Endovascular Oncology
Other Study IDs: ILI01; ILI100513 (Other: IGEVO)
Record Dates: First submitted 2013-08-06; First posted 2013-08-12 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Melanoma
Keywords: Isolated limb infusion; Melphalan; Limb Melanoma; Tumor response
MeSH Terms: conditions — Melanoma | interventions — Melphalan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Melphalan: Day +1:
  Intra femoral infusion of Melphalan at the dosage 1mg/ Kg
  Intra femoral infusion of Melphalan Second ILI treatment can be repeated at side effects recovery ( following oncologist ' s planning of cure).
  Day +30: The above procedure is repeated.
  Day +90: In case of response, a third administration following the above procedures will be repeated.
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Melphalan — Melphalan 1mg/kgr is rapidly infused into the isolated limb via the arterial catheter after the inflation of venous baloon catheter.
  Other Names: Alkeran

SUMMARY:
In-transit metastases occur in approximately 3% of melanoma patients, can be very symptomatic and the survival in this group may be prolonged. In-transit melanoma metastases are often confined to a limb. In this circumstance, treatment by isolated limb perfusion or isolated limb infusion can be a remarkably effective regional treatment option. Isolated limb infusion (ILI) was introduced in 1992 and is a technique used to deliver regional chemotherapy to treat advanced melanoma confined to a limb. Regional chemotherapy with melphalan delivered by isolated limb perfusion (ILP) or ILI are effective treatment options for in-transit melanoma and are generally well tolerated.

ILI is a less invasive and simpler alternative to ILP. Complete response rates are 45- 69% for ILP and 23-44% for ILI. The limb is often warmed to lower temperatures in ILI compared to ILP and the limb becomes progressively more hypoxic and acidotic during ILI, each of these parameters potentially having an effect on outcome. ILP & ILI are used primarily as palliative options when excision of in-transit metastases is unfeasible but can be used as an adjunctive procedure to surgery, for other tumour types such as merkel cell carcinoma, and can be repeated if indicated. For ILI correction of melphalan dose for ideal body weight has been shown to substantially decrease the rates of severe local toxicity while maintaining complete response rates, but overall response rate is reduced.

Response to ILI, moreover, is different in upper and lower limbs. ILI for Upper limbs disease is associated with similar complete response rates but lower toxicity than ILI for Lower limbs E disease and with different physiologic sequelae despite comparable methods. The Upper limbs appears relatively resistant to toxic effects of melphalan-based ILI as currently performed, which suggests a potential for further optimization of drug dosing for Upper limbs ILI.

Regional therapy is an excellent therapeutic modality for disease limited to a limb and furthermore serves as an excellent model for scientific investigation, both clinical and translational. In this study we want to collect data on isolated limb infusion of chemotherapy to monitor efficacy and tolerability in patients with melanoma metastases of the arm or leg that cannot be removed by surgery.

DETAILED DESCRIPTION:
This is an observational study and the treatment is related to the experiences and economical availability of each center.

Study Design: Prospective observational study . Primary objective: To collect data on tumor response and progression free survival after administration of melphalan.

Secondary objectives: To collect data on survival rate, time to progression, morbidity tolerability of treatment, number of treatment required to achieve objective response and improvement of quality of life (Edmonton questionnaire)

Treatment under observation :

Patients undergo fluoroscopic placement of angiographic arterial and venous catheters into the appropriate extremity in order to infuse the drug (artery) and to stop the out flow (venous with balloon catheter). Melphalan 1mg/kgr is rapidly infused into the isolated limb via the arterial catheter after the inflation of venous balloon catheter. Then the circulation of the limb is blocked with a pneumatic cuff at the root of the limb . Patients with little or no response at 8 weeks may receive up to 2 additional treatments at the discretion of the treating physician.

Patients are followed at 1-2 weeks, 3-4 weeks, 6-8 weeks, and then every 3-6 months thereafter as deemed necessary by the treating physician.

Day -1 Melphalan 1mg/ Kgr has been prepared at Pharmacy.

Day 0: prehydration, antibiotic prophylaxis and setting up of a therapeutic scheme appropriate for analgesic prophylaxis (3-day duration) as previously reported (25)

Day +1:

Upon admittance to the radiology room, 1 vial of tropisetron (diluted in 100ml of physiological solution) administered by slow drip.

During infusion of the Melphalan into the artery, 1 vial of morphine hydrochloride diluted in 100 ml i.v. to be repeated one hour after the procedure and if necessary also after 6 hours.

Tropisetron i.v. if needed. Intra-arterial premedication with 1 vial of verapamil diluted in 4 ml of normal saline solution followed by 4 ml of lidocaine.

Intra femoral infusion of Melphalan Second ILI treatment could be repeated at side effects recovery ( following oncologist ' s planning of cure).

Day +30: The above procedure is repeated.

Day +90: In case of response, a third administration following the above procedures will be repeated.

Evaluation of response:

Response must be assessed by repeating the following examinations at Day 30, Day 90 and Day 120 after start of treatment:

Limb-Chest-abdomen CAT scan with and without contrast medium (refer to Section 4). Evaluation will be based on Response Evaluation Criteria in Solid Tumors (RECIST ) criteria [20-24 ] cancer markers (CEA, cancer antigen (CA) 19.9)

Assessment of quality of life The Edmonton Symptom Assessment System (ESAS) is used to monitor health conditions and quality of life.

Assessment of quality of life is performed during the baseline visit and at Day 30, Day 60 and Day 120 from start of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven primary or recurrent, regional melanoma or soft tissue sarcoma that is not amenable to surgical resection
2. Majority (greater than 95%) of disease must be distal to the apex of the femoral triangle in the lower limb and the deltoid insertion in the upper limb
3. Bidimensionally measurable disease in the extremity
4. Patients with disease beyond the limb are eligible if their extremity disease requires palliative treatment in the judgment of their physician
5. Age: more than 18
6. Karnofsky 70-100%
7. Life expectancy: At least 6 months
8. Hematopoietic: WBC at least 3,000/mm^3
9. Renal: Creatinine less than 2.0 mg/dL
10. At least 4 weeks since prior antitumor therapy and recovered
11. At least 2 weeks since prior antibiotics

Exclusion Criteria:

1. Signs or symptoms of vascular insufficiency (no history of claudication or other ischemic peripheral vascular disease)
2. pregnant or nursing
3. other concurrent serious illness
4. severe diabetes
5. prior extremity complications due to diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-07; Primary Completion 2019-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Tumor response | 12 months
  Response must be assessed by repeating the following examinations, at Day 30, Day 90 and Day 120 after start of treatment:
  Chest-abdomen CAT scan with and without contrast medium (refer to Section 4). Evaluation will be based on RECIST criteria [18-22 ] cancer markers (CEA, CA 19.9)

SECONDARY OUTCOMES:
survival rate | 12 months
  percentage of patients alive
time to progression | 12 months
  time from treatment start to progression
number of adverse events | 4 months
  number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Giammaria Fiorentini, MD, Principal Investigator — International Group of Endovascular Oncology
Locations (1):
- Azienda Ospedaliera Ospedali Riuniti Marche Nord, Presidio Ospedaliero San Salvatore, Pesaro, PU, Italy

REFERENCES:
- [Result] Ruscitti C, Guadagni S, Russo F, Palumbo G, Fiorentini G, Mambrini A, Cantore M, Kanavos E, Pinto A, Amicucci G. Thoracic stop-flow perfusion for refractory lymphoma: a phase I-II evaluation trial. In Vivo. 2009 May-Jun;23(3):447-57. PMID 19454513
- [Result] Guadagni S, Clementi M, Valenti M, Fiorentini G, Cantore M, Kanavos E, Amicucci G. Thoracic stop-flow perfusion in the treatment of refractory malignant pleural mesothelioma: a phase I-II evaluation/trial. In Vivo. 2006 Nov-Dec;20(6A):715-8. PMID 17203752
- [Result] Guadagni S, Santinami M, Patuzzo R, Pilati PL, Miotto D, Deraco M, Rossi CR, Fiorentini G, Di Filippo F, Valenti M, Amicucci G. Hypoxic pelvic and limb perfusion with melphalan and mitomycin C for recurrent limb melanoma: a pilot study. Melanoma Res. 2003 Feb;13(1):51-8. doi: 10.1097/00008390-200302000-00009. PMID 12569285
- [Result] Guadagni S, Russo F, Rossi CR, Pilati PL, Miotto D, Fiorentini G, Deraco M, Santinami M, Palumbo G, Valenti M, Amicucci G. Deliberate hypoxic pelvic and limb chemoperfusion in the treatment of recurrent melanoma. Am J Surg. 2002 Jan;183(1):28-36. doi: 10.1016/s0002-9610(01)00841-8. PMID 11869699
- [Derived] Guadagni S, Zoras O, Fiorentini G, Masedu F, Lasithiotakis K, Sarti D, Farina AR, Mackay AR, Clementi M. A Prospective Study of Intraarterial Infusion Chemotherapy in Advanced Wild-Type BRAF Melanoma Patients. J Surg Res. 2021 Dec;268:737-747. doi: 10.1016/j.jss.2021.05.054. Epub 2021 Jul 10. PMID 34253376
- [Derived] Guadagni S, Fiorentini G, Papasotiriou I, Apostolou P, Masedu F, Sarti D, Farina AR, Mackay AR, Clementi M. Circulating tumour cell liquid biopsy in selecting therapy for recurrent cutaneous melanoma with locoregional pelvic metastases: a pilot study. BMC Res Notes. 2020 Mar 24;13(1):176. doi: 10.1186/s13104-020-05021-5. PMID 32204733
- [Derived] Guadagni S, Palumbo G, Fiorentini G, Clementi M, Marsili L, Giordano AV, Masedu F, Valenti M. Surgical versus percutaneous isolated pelvic perfusion (IPP) for advanced melanoma: comparison in terms of melphalan pharmacokinetic pelvic bio-availability. BMC Res Notes. 2017 Aug 15;10(1):411. doi: 10.1186/s13104-017-2738-y. PMID 28810925
- See also: International group of endovascular oncology (IGEVO) website — http://igevo.jimdo.com/